CLINICAL TRIAL: NCT05856019
Title: Effects of J Stroke Myofascial Release on Plantar Fascia Versus Ischemic Release on Gastrocnemius in Patients With Planter Fasciitis
Brief Title: Effects of J Stroke Myofascial Release in Patients With Planter Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0122
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Plantar Fascitis
Keywords: planter fascitis; J stroke myofascial release; Ischemic release on gastrocnemius

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- J Stroke Myofascial Release (Experimental): Patient is in prone lying position with foot supported. Pressure is applied with the heel of the opposite hand, while a stroke in the shape of the letter J is applied in the direction of the restriction, with two or three fingers, which creates some torque at the end. Myofascial Release techniques will be performed for 20 repetitions.
  Interventions: Other: J Stroke Myofascial Release
- Ischemic Release on Gastrocnemius through Dry Cupping (Active Comparator): Dry cupping will provided to the subjects thrice a week for 4 weeks in the dry cupping therapy group, a plastic cupping bell will be used. Cups will applied to the painful site for 10 minutes in each session. A manual hand pump was used to create the vacuum for suction. The intensity of the vacuum will based on subject tolerance.
  Interventions: Other: Ischemic Release on Gastrocnemius through Dry Cupping

INTERVENTIONS:
Other: J Stroke Myofascial Release — Group A will receive J stroke myofascial release on planter fascia (with hot pack for 10-15 minutes on calf) 3 sessions per week for 4 weeks.
  Arms: J Stroke Myofascial Release
Other: Ischemic Release on Gastrocnemius through Dry Cupping — Group B will ischemic release on gastrocnemius (with hot pack for 10-15 minutes on calf) 3 sessions per week for 4 weeks.
  Arms: Ischemic Release on Gastrocnemius through Dry Cupping

SUMMARY:
The purpose of the study is to compare the effects of j stroke myofascial release on planter fascia versus ischemic release on gastrocnemius in patients with planter fasciitis.

DETAILED DESCRIPTION:
Planter fasciitis is commonly occur in athletes and females who wear flat shoes. It is caused by the loss of planter fascia flexibility that leads to mechanical overloading of fascial structures. There are some risk factors that are important to consider include age, leg length difference, inadequate footwear, inappropriate walking and running patterns and increased planter fascia thickness. Planter fascia thickness more than 4mm can be considered as an indicative of planter fasciitis.

Myofascial soft tissue mobilization is a low load, long duration stretch to the myofascial complex technique that is given in both acute and chronic conditions which in caused by tightness and soft tissue restriction in the patients with planter fasciitis to restore length, decrease pain and to improve function.

Cupping therapy on gastrocnemius is a medical technique that applies negative pressure over pain areas and pressure points that alleviates pain and improve blood circulation. it could be low-cost and convenient alternative technique to treat planter fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60years
* Both Genders
* Chronic pain
* Heel pain with current and previous diagnosis of planter faucitis
* Unilateral planter fascia involvement
* Mild to moderate heel pain with NPRS pain score value between 2-6

Exclusion Criteria:

* Recent surgery to ankle joint
* Impaired sensations
* Open wound
* Peripheral vascular disease
* Recent fractures (<6 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
NPRS | 1st day, 2nd week, 4th week
  Numeric Rating Scale (NPRS) is most frequently used instruments to measure the intensity of ankle pain with an 11-point numerical pain rating scale (NPRS), where 0 is the absence of pain and 10 represents maximum pain. 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs).

SECONDARY OUTCOMES:
FFI | 1st day, 2nd week, 4th week
  A Foot Function Index (FFI) was developed to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales. The FFI should prove useful for both clinical and research purposes
Goniometer | 1st day, 2nd week, 4th week
  Goniometers are commonly used to determine ROM of the ankle joint. Goniometers are considered valid and reliable clinical tools for assessing range of motion of joints of the extremities

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, phd, Principal Investigator — Riphah International University
Locations (1):
- Ortho-Med Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akter S, Hossain MS, Hossain KMA, Uddin Z, Hossain MA, Alom F, Kabir MF, Walton LM, Raigangar V. Comparison of Structural Diagnosis and Management (SDM) approach and MyoFascial Release (MFR) for improving plantar heel pain, ankle range of motion and disability: A randomized clinical trial. J Man Manip Ther. 2024 Aug;32(4):368-377. doi: 10.1080/10669817.2023.2214020. Epub 2023 May 24. PMID 37222021
- [Background] Karagounis P, Tsironi M, Prionas G, Tsiganos G, Baltopoulos P. Treatment of plantar fasciitis in recreational athletes: two different therapeutic protocols. Foot Ankle Spec. 2011 Aug;4(4):226-34. doi: 10.1177/1938640011407320. PMID 21868796
- [Background] Malik S, Anand P, Bhati P, Hussain ME. Effects of dry cupping therapy on pain, dynamic balance and functional performance in young female with recreational runners chronic plantar fasciitis. Sports Orthopaedics and Traumatology. 2022;38(2):159-70.
- [Background] Tamboli U, Patil C. Effect of myofascial release with lower limb strengthening on plantar fasciitis. International Journal of Physical Education, Sports and Health. 2021;8(1):27-31.
- [Background] Vijayakumar M, Jaideep A, Khankal R, Gazbare P, Abraham B. Effectiveness of compressive myofascial release vs instrument assisted soft tissue mobilization in subjects with active trigger points of the calf muscle limiting ankle dorsiflexion. Int J Health Sci Res. 2019;9(4):98-106.
- [Background] Farooq N, Aslam S, Bashir N, Awan WA, Shah M, Irshad A. Effectiveness of transverse friction massage of Flexor digitorum brevis and Calf muscle stretching in Plantar fasciitis on foot function index scale: A randomized control trial. Isra Med J. 2019;1(4):305-9.
- [Background] Prakash S, Misra A. Effect of manual therapy versus conventional therapy in patients with plantar fasciitis-a comparative study. Int J Physiother Res. 2014;2(1):378-82.
- [Background] Armagan Alpturker K, Cerrahoglu ABL, Orguc IS. Evaluation Effects of Laser Therapy and Extracorporeal Shock Wave Therapy with Clinical Parameters and Magnetic Resonance Imaging for Treatment of Plantar Fasciitis in Patients with Spondyloarthritis: A Randomized Controlled Trial. Int J Rheumatol. 2020 Aug 27;2020:4386361. doi: 10.1155/2020/4386361. eCollection 2020. PMID 32908536